CLINICAL TRIAL: NCT00097630
Title: Cognitive Impairment in the ICU: Evaluation and Outcomes
Brief Title: ABC Trial: Awakening and Breathing Controlled
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: St. Thomas Foundation, Tennessee (Other); Vanderbilt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0011; 5K23AG001023-04 (NIH)
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2008-08

CONDITIONS: Aging; Respiration, Artificial
Keywords: mechanical ventilation; delirium; sedation scoring; cognitive impairment; ventilation weaning
MeSH Terms: conditions — Respiratory Aspiration; Delirium; Cognitive Dysfunction

INTERVENTIONS:
Procedure: SAT: Spontaneous Awakening Trial
Procedure: SBT: Spontaneous Breathing Trial

SUMMARY:
The purpose of this study is to determine the impact of a new RN/RRT (Registered Nurse/Registered Respiratory Therapist) directed 2-step protocol to wean patients off of a ventilator. This protocol involves daily attempts to halt sedation (spontaneous awakening trials) combined with daily assessments of patients while they are breathing on their own (spontaneous breathing trials).

DETAILED DESCRIPTION:
Unnecessary delays in removing patients from mechanical ventilation increase morbidity, mortality, and cost. According to recently published guidelines, the current standard of care for weaning involves the daily assessment of patients while they are breathing spontaneously, also known as spontaneous breathing trials (SBT). While there are important data to support a daily cessation of sedatives and analgesics to the point of patient awakening, the benefit of combining such a daily spontaneous awakening trial (SAT) and an SBT is not known.

This multi-center, randomized controlled trial will test whether a 2-step process of weaning that combines a daily awakening trial (achieved by stopping all sedatives and narcotics every morning) with a daily spontaneous breathing trial is superior to the current standard of care.

The number of days the patient is able to live off the ventilator is the primary question being studied. The secondary questions include the number of days the patient is in Intensive Care Unit (ICU) and the hospital, the complications associated with being on the ventilator (such as the duration and severity of delirium and coma), and in-hospital and one-year mortality. Also, cognitive, psychological, and functional/quality of life outcomes will be measured at discharge and 3 and 12 months later.

In addition, the study will measure plasma drug levels twice daily on five sequential days within 30 minutes of testing with highly reliable and well validated instruments to measure sedation level (i.e., RASS) and delirium (i.e. CAM-ICU).

ELIGIBILITY:
Inclusion Criteria:

* Recently on mechanical ventilation (less than 2 weeks prior to enrollment)
* Require mechanical ventilation for more than 12 hours
* Over 18 years old
* Under the services of medicine, cardiology, and neurology

Exclusion Criteria:

* Admission after cardiopulmonary arrest
* Inability to obtain informed consent
* Existence of an extubation order at the time of the evaluation
* Dependence upon mechanical ventilation for 2 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334
Dates: Start 2003-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Ventilator free days

SECONDARY OUTCOMES:
Length of stay in the ICU and hospital
28-day and 1-year survival
Duration of coma and delirium
Cognitive function | at discharge, 3 months, and 12 months
Psychological status | at discharge, 3 months, and 12 months
Functional status | at discharge, 3 months, and 12 months
Quality of life | at discharge, 3 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: E Wesley Ely, MD, MPH, Principal Investigator — Vanderbilt University Medical Center; Brenda T Pun, RN, ACNP, Study Director — Vanderbilt University Medical Center; Richard W Light, MD, Principal Investigator — St. Thomas Hospital
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania - Presbyterian Medical Center, Philadelphia, Pennsylvania
  - St. Thomas Hospital, Nashville, Tennessee

REFERENCES:
- [Background] Ely EW, Baker AM, Dunagan DP, Burke HL, Smith AC, Kelly PT, Johnson MM, Browder RW, Bowton DL, Haponik EF. Effect on the duration of mechanical ventilation of identifying patients capable of breathing spontaneously. N Engl J Med. 1996 Dec 19;335(25):1864-9. doi: 10.1056/NEJM199612193352502. PMID 8948561
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Result] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Derived] Jackson JC, Girard TD, Gordon SM, Thompson JL, Shintani AK, Thomason JW, Pun BT, Canonico AE, Dunn JG, Bernard GR, Dittus RS, Ely EW. Long-term cognitive and psychological outcomes in the awakening and breathing controlled trial. Am J Respir Crit Care Med. 2010 Jul 15;182(2):183-91. doi: 10.1164/rccm.200903-0442OC. Epub 2010 Mar 18. PMID 20299535
- See also: Focus on delirium and other issues associated with ICU patients. — http://www.ICUdelirium.org